CLINICAL TRIAL: NCT02708563
Title: Meconium Aspiration Syndrome and Non-vigorous Neonates-Pilot Study
Brief Title: Meconium Aspiration and Tracheal Suctioning-Feasibility Study
Acronym: MATS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Inadequate funds allocated for study completion
Sponsor: St. Louis University (Other)
Collaborators: American Academy of Pediatrics (Other)
Responsible Party: Principal Investigator, Marya Strand, MD, Associate Professor of Pediatrics, St. Louis University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SLU-19817
Record Dates: First submitted 2016-03-02; First posted 2016-03-15 (Estimated); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Meconium Aspiration Syndrome
Keywords: meconium; neonatal resuscitation
MeSH Terms: conditions — Meconium Aspiration Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate intubation (Experimental): These infants will have immediate endotracheal suctioning after delivery. They will then have resuscitation per Neonatal Resuscitation Program guidelines.
  Interventions: Procedure: Immediate intubation
- Immediate resuscitation (Experimental): These infants will have immediate resuscitation per the Neonatal Resuscitation Program guidelines without endotracheal suctioning.
  Interventions: Procedure: Immediate resuscitation

INTERVENTIONS:
Procedure: Immediate intubation — Infants that are not vigorous at delivery will receive immediate tracheal suctioning
  Arms: Immediate intubation
Procedure: Immediate resuscitation — Infants that are not vigorous at delivery will receive immediate initial steps of resuscitation and PPV if needed
  Arms: Immediate resuscitation

SUMMARY:
Feasibility study to randomize non-vigorous newborn infants born through meconium-stained amniotic fluid to endotracheal suctioning or immediate resuscitation.

DETAILED DESCRIPTION:
This will be a pilot feasibility trial of endotracheal intubation and suctioning versus routine resuscitation for term, non-vigorous newborns born through meconium-stained amniotic fluid to compare the incidence of meconium aspiration syndrome, extracorporeal membrane oxygenation or death.

ELIGIBILITY:
Inclusion Criteria:

* Term newborns (>37 weeks of gestation)
* Delivery through meconium-stained amniotic fluid
* Mothers >18 years of age

Exclusion Criteria:

* No consent from mother
* Infant vigor at delivery (muscle tone and respiratory effort)
* Prenatally diagnosed major anomalies (excluding gastroschisis)
* Plan to not resuscitate infant
* Family does not speak English

Max Age: 5 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2019-07 (Estimated); Primary Completion 2020-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Ability to identify, consent, enroll and randomize 70% of eligible infants into study. | 18 months
  Feasibility measures
The number of infants in the study who develop meconium aspiration syndrome, require extracorporeal membrane oxygenation or die | 18 months
  Clinical outcome measure

IPD SHARING:
Plan to Share IPD: No